CLINICAL TRIAL: NCT07221253
Title: Phase III, Randomized, Open-label, Global, Multicenter Study of Rilvegostomig or Durvalumab in Combination With Chemotherapy as a First-line Treatment for Patients With Advanced Biliary Tract Cancer (ARTEMIDE-Biliary02)
Brief Title: A Study of Rilvegostomig or Durvalumab Plus Chemotherapy for First-Line Treatment of Biliary Tract Cancer (ARTEMIDE-Biliary02)
Acronym: AB02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D702NC00001
Record Dates: First submitted 2025-10-01; First posted 2025-10-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Biliary Tract Cancer
Keywords: Rilvegostomig; Durvalumab; Biliary Tract Cancer; Bispecific Antibody; PD-L1; TIGIT; Initially Unresectable; Recurrent; Intra-hepatic cholangiocarcinoma; Extra-hepatic cholangiocarcinoma; Gallbladder cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Recurrence; Gallbladder Neoplasms | interventions — durvalumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Durvalumab IV infusion + chemotherapy combination (Gemcitabine/Cisplatin)
  Interventions: Drug: Durvalumab; Drug: Gemcitabine/Cisplatin
- Experimental Arm (Experimental): Rilvegostomig IV infusion + chemotherapy combination (Gemcitabine/Cisplatin)
  Interventions: Drug: Rilvegostomig; Drug: Gemcitabine/Cisplatin

INTERVENTIONS:
Drug: Rilvegostomig — Rilvegostomig IV (intravenous) Q3W
  Other Names: AZD2936
  Arms: Experimental Arm
Drug: Durvalumab — Durvalumab 1500mg IV (intravenous) Q3W for up to 8 cycles (21days). Then Q4W.
  Other Names: IMFINZI
  Arms: Control Arm
Drug: Gemcitabine/Cisplatin — Gemcitabine/Cisplatin IV (Intravenous) 1000 mg/m2 plus cisplatin 25 mg/m2 on Day 1 and Day 8 of each 21-day cycle

SUMMARY:
The purpose of this study is to measure the efficacy and safety of rilvegostomig with gemcitabine plus cisplatin vs. durvalumab with gemcitabine plus cisplatin as first line treatment for patients with advanced BTC.

ELIGIBILITY:
Key inclusion Criteria:

* Histologically confirmed adenocarcinoma of the biliary tract, including intra-hepatic or extra-hepatic cholangiocarcinoma (CCA) and gallbladder carcinoma (GBC).
* Unresectable locally advanced or metastatic BTC, previously untreated in the advanced disease setting
* Known PD-L1 status assessed at a central laboratory using an acceptable tumor sample.
* Measurable disease by RECIST 1.1 criteria using CT or MRI and is suitable for accurate repeated measurements.
* ECOG Performance Status of 0 or 1 with no deterioration (ie, ECOG PS > 1) over the previous 2 weeks prior to baseline at screening and prior to randomization.
* Adequate bone marrow and organ function.

Key exclusion Criteria:

* Ampullary carcinoma
* Any prior systemic therapy received for unresectable, locally advanced or metastatic BTC.
* Any prior exposure to any other therapy targeting immune-regulatory receptors or mechanisms.
* Any concurrent chemotherapy, radiotherapy, immunotherapy, investigational, biologic, or hormonal therapy for cancer treatment other than those under investigation in this study.
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* Active or ongoing interstitial lung disease/pneumonitis (of any grade), serious chronic gastrointestinal conditions associated with diarrhea, or active non-infectious skin disease (including any grade rash, urticaria, dermatitis, ulceration, or psoriasis) requiring systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2029-07-04 (Estimated); Study Completion 2029-07-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in the PDL1 ≥ 1% population | approximately 4 years
  Overall Survival is defined as time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Overall Survival in the intent to treat (ITT) population | approximately 4 years
  Overall Survival is defined as time from randomization until the date of death due to any cause.
Progression Free Survival (PFS) in the PDL1 ≥ 1% population | approximately 4 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1, or death due to any cause (in the absence of progression), whichever occurs first.
Progression Free Survival (PFS) in the intent to treat (ITT) population | approximately 4 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1 or death due to any cause (in the absence of progression), whichever occurs first.
Objective Response Rate (ORR) in the PDL1 ≥ 1% population | approximately 4 years
  ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR using RECIST 1.1.
Objective Response Rate (ORR) in the intent to treat (ITT) population | approximately 4 years
  ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR using RECIST 1.1.
Duration of Response (DoR) in the PDL1 ≥ 1% population | approximately 4 years
  DoR is defined as the time from the date of first documented response until the date of documented progression using RECIST 1.1 or death due to any cause (in the absence of progression), whichever occurs first.
Duration of Response (DoR) in the intent to treat (ITT) population | approximately 4 years
  DoR is defined as the time from the date of first documented response until the date of documented progression using RECIST 1.1 or death due to any cause (in the absence of progression), whichever occurs first.
Time to Second Progression or death (PFS2) in the PDL1 ≥ 1% population | approximately 4 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial progression event), after the start of the first subsequent therapy, or death from any cause, whichever occurs first.
Time to Second Progression or death (PFS2) in the intent to treat (ITT) population | approximately 4 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial progression event), after the start of the first subsequent therapy, or death from any cause, whichever occurs first.
Assess the safety and tolerability of rilvegostomig in combination with chemotherapy vs durvalumab in combination with chemotherapy | approximately 4 years
  Safety and tolerability will be evaluated by the proportion of treated patients with occurrence of AEs and SAEs as assessed by CTCAE v5.0.
Immunogenicity of Rilvegostomig | approximately 4 years
  Presence of ADA for rilvegostomig (confirmatory results, titres and neutralising antibodies for confirmed positive samples).
PK of rilvegostomig: Lowest observed concentration of study drug before the next dose is administered (Ctrough) | Up to 12 weeks after disease progression
  Lowest observed plasma concentration of the study drug (Ctrough) prior to next dose
PK of rilvegostomig: Maximum plasma concentration of the study drug (Cmax) | Up to 12 weeks after disease progression
  Maximum observed plasma concentration of rilvegostomig
Serum rilvegostomig concentration | Up to 12 weeks after disease progression
  To assess drug exposure (serum concentration) of IV rilvegostomig.
Assess patient reported biliary tract cancer symptoms (pain) | Up to 12 weeks post disease progression
  Patient reported biliary tract cancer symptoms (pain) will be evaluated by the proportion of randomized patients with maintained or improved pain as assessed by the EORTC Item Library 445 and EORTC Item Library 446 (custom questionnaires that include measures of pain-in back, in stomach area, during the night; min/max values from 1-4, with higher scores indicating a worse outcome).
Assess patient reported global health status/quality of life (GHS/QoL) | Up to 12 weeks post disease progression
  Patient reported GHS/QoL will be evaluated by the proportion of randomized patients with maintained or improved GHS/QoL as assessed by the EORTC Item Library 172 (custom questionnaire that includes measures of overall health and overall quality of life; min/max values from 1-7, with higher scores indicating a better outcome).

CONTACTS AND LOCATIONS:
Locations (144):
- United States (27):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Duarte, California
  - Research Site, Orange, California
  - Research Site, Santa Monica, California
  - Research Site, Stanford, California
  - Research Site, Aurora, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Santa Fe, New Mexico
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Sioux Falls, South Dakota
- Australia (2):
  - Research Site, Darlinghurst
  - Research Site, Murdoch
- Belgium (5):
  - Research Site, Anderlecht
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (19):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Lishui
  - Research Site, Luoyang
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Weifang
  - Research Site, Wuhan
  - Research Site, Xi'an
- France (4):
  - Research Site, Clichy
  - Research Site, Grenoble
  - Research Site, Marseille
  - Research Site, Vandœuvre-lès-Nancy
- Germany (14):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Karlsruhe
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Ulm
- India (5):
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Kolhāpur
  - Research Site, Mumbai
  - Research Site, Surat
- Italy (5):
  - Research Site, Castellana Grotte
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Rome
  - Research Site, Rozzano
- Japan (11):
  - Research Site, Chiba
  - Research Site, Kashiwa
  - Research Site, Kawasaki-shi
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Suita-shi
  - Research Site, Takatsuki-shi
  - Research Site, Ube
  - Research Site, Yokohama
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Utrecht
- Poland (5):
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Warsaw
- South Korea (4):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Santander
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Ongkharak
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Erzurum
  - Research Site, Istanbul
  - Research Site, Konya
  - Research Site, Seyhan
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, Greater London
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure